CLINICAL TRIAL: NCT00005013
Title: A Placebo Controlled Clinical Trial of a Standardized Extract of Hypericum Perforatum in Major Depressive Disorder
Brief Title: Treatment of Major Depression With St. John's Wort (Hypericum)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: N01 MH70007; DSIR CT
Record Dates: First submitted 2000-03-31; First posted 2000-04-03 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2006-03

CONDITIONS: Major Depression
Keywords: Antidepressive Agents; Depression; Depressive Disorder; Herbs; Hypericum; Medicine, Herbal; Plant Extracts; Alternative Medicine
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — Sertraline; Hypericum extract LI 160

INTERVENTIONS:
Drug: Sertraline
Drug: Hypericum perforatum (St. John's wort)

SUMMARY:
The purpose of this trial is to study the acute efficacy and safety of a standardized extract of the herb Hypericum perforatum (St. John's Wort), called hypericum for purposes of this trial, in the treatment of patients with major depression.

Clinical depression is a serious medical disorder that can be debilitating and can lead to suicide. There is growing public interest in claims that hypericum may be an effective treatment for depression. Although it is widely prescribed in Europe, no studies of its long-term use have been conducted, and published studies have treated different types of patients and have used several different doses. The toxicity and side effects of hypericum appear to be substantially less than those of standard tricyclic antidepressant medications, and thus hypericum may be more acceptable to patients. In addition, the cost is significantly less than standard antidepressant medications. Published studies assessed acute efficacy and lasted between 4 and 12 weeks (most being 4-6 weeks). The longer-term effects of hypericum have not been evaluated. There is a need for a large-scale, controlled clinical trial to assess whether Hypericum has a significant therapeutic effect in patients with clinical depression.

Patients are assigned randomly (like tossing a coin) to receive St. John's wort, Sertraline (Zoloft), or a placebo (sugar pill) for 8 weeks. This is a double-blind study, meaning neither the patient nor the doctor will know which treatment is being assigned. Patients who respond well to the treatment will continue on the assigned treatment for an additional 4 months. Patients will have regular follow-up visits to monitor their symptoms and any side effects they experience.

DETAILED DESCRIPTION:
This trial will determine the acute antidepressant efficacy of a standardized extract of hypericum (St. John's Wort) for the treatment of major depressive disorder.

For this trial, the primary efficacy analysis will be evaluated at 8 weeks. For observational purposes, a 4-month double blind continuation (6 months total treatment) in treatment responders would enable an approximation of the effectiveness of maintenance treatment with this medication. No published studies have included a selective serotonin re-uptake inhibitor (SSRI) comparator. While this trial will not compare the efficacy of hypericum to an SSRI, having an SSRI arm of sertraline (Zoloft) will allow an evaluation of the validity of the trial.

336 eligible patients will be randomly assigned to double-blind treatment with hypericum, sertraline, or placebo following a one-week placebo lead-in period (between screening and baseline). All treatment groups will consist of 112 patients and will be followed for an eight-week period. Treatment responders will be continued on the randomly assigned treatment arm for an additional 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Major depression assessed by Structured Clinical Interview for DSM-IV Axis I Disorders (SCID; First et al, 1995)
* Minimum score greater than or equal to 20 on the 17-item Hamilton Depression (HAM-D) Scale at screen and at baseline
* GAF of 60 or less (moderate symptoms) at screen and at baseline
* HAM-D cannot decrease by 25% or more between screening and baseline
* Capacity to give informed consent and to follow study procedures.
* Abstinence or effective method of contraception throughout the study

Exclusion Criteria:

* Scores greater than 2 on the "suicide" item of HAM-D, or history of suicide attempt(s) in the past 12 months
* Current suicidal or homicidal risk, as determined by the investigator
* Women of childbearing age who are pregnant, planning pregnancy in the next 6 months, breast-feeding, or not using medically acceptable means of birth control (hormonal treatment such as birth control pill, injection or implant, IUD, or double barrier of condom and diaphragm together is acceptable; primary use of condom, sponge or diaphragm alone (single barrier) is not acceptable because these may carry a higher rate of failure when used alone
* Clinically significant liver disease (such as hepatitis, cirrhosis, etc); or clinically significant elevation of liver enzyme tests (two times the upper limit of normal; asymptomatic Gilbert's syndrome is not an exclusion). 4. Serious or unstable medical illness. 5. History of seizure disorder (other than febrile).
* Any of the following DSM-IV diagnoses by SCID: current (within past 6 months) alcohol or other substance abuse disorder; schizophrenia, schizo-affective, or other psychotic disorder; bipolar disorder; current panic disorder or obsessive compulsive disorder; history of psychotic features of affective disorder (mood congruent or incongruent)
* Clinical or laboratory evidence of untreated or unstable thyroid disorder
* Failed to respond to at least two adequate antidepressant trials (defined as 6 weeks or more treatment with either greater than or equal to 150 mg imipramine, or tricyclic equivalent), or greater than or equal to 60 mg of phenelzine, or MAOI equivalent, or greater than or equal to 100 mg of sertraline, or its SSRI equivalent
* Have taken sertraline or any form of hypericum during this current episode of depression at any dose level, daily, for at least one month, within the past 6 months
* Current (within past 6 months) use of other prescription or non-prescription drugs, including anticonvulsants and other medications with significant psychotropic properties, antiretroviral medications, cyclosporine, digoxin, coumadin, dietary supplements, natural remedies, and botanical preparations (eg, hypericum, kava, valerian)
* Have had other investigational drugs within 30 days or other psychotropic medication within 21 days of baseline (6 weeks for fluoxetine)
* Known allergy or hypersensitivity to the study medications
* Positive drug urine screen
* Have been in psychotherapy for 2 months or less at the time of enrollment into the study
* Receiving psychotherapies which are specifically designed to treat depression, eg, interpersonal psychotherapy during the study period
* Mental retardation or cognitive impairment, or any disorder that might interfere with their ability to consent or follow study procedures and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-12; Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Davidson, Principal Investigator — Duke Univ Med Ctr
Locations (12):
- United States (12):
  - Feighner Research Institute, San Diego, California
  - Stanford Univ School of Medicine, Stanford, California
  - Harbor-UCLA Rsch and Education Inst, Torrance, California
  - Univ of South Florida College of Med, Tampa, Florida
  - Emory Mood and Anxiety Disorders Clinical Trials Program, Atlanta, Georgia
  - McLean Hospital, Belmont, Massachusetts
  - Eastside Comprehensive Medical Services, New York, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati Medical Ctr, Cincinnati, Ohio
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Seattle Clinical Research Center, Seattle, Washington
  - Dean Foundation for Hlth Rsch and Education, Middleton, Wisconsin

REFERENCES:
- [Result] Hypericum Depression Trial Study Group; Davidson JR, Gadde KM, Fairbank JA, Krishnan KRR, Califf RM, Binanay C, Parker CB, Pugh N, Hartwell TD, Vitiello B, Ritz L, Severe J, Cole JO, de Battista C, Doraiswamy PM, Feighner JP, Keck P, Kelsey J, Lin KM, Londborg PD, Nemeroff CB, Schatzberg AF, Sheehan DV, Srivastava RK, Taylor L, Trivedi MH, Weisler RH. Effect of Hypericum perforatum (St John's wort) in major depressive disorder: a randomized controlled trial. JAMA. 2002 Apr 10;287(14):1807-14. doi: 10.1001/jama.287.14.1807. PMID 11939866
- [Result] Vitiello B, Shader RI, Parker CB, Ritz L, Harlan W, Greenblatt DJ, Gadde KM, Krishnan KR, Davidson JR. Hyperforin plasma level as a marker of treatment adherence in the National Institutes of Health Hypericum Depression Trial. J Clin Psychopharmacol. 2005 Jun;25(3):243-9. doi: 10.1097/01.jcp.0000162801.72002.85. PMID 15876903
- [Derived] Chen JA, Vijapura S, Papakostas GI, Parkin SR, Kim DJ, Cusin C, Baer L, Clain AJ, Fava M, Mischoulon D. Association between physician beliefs regarding assigned treatment and clinical response: re-analysis of data from the Hypericum Depression Trial Study Group. Asian J Psychiatr. 2015 Feb;13:23-9. doi: 10.1016/j.ajp.2014.12.002. Epub 2014 Dec 9. PMID 25544195
- [Derived] Grobler AC, Matthews G, Molenberghs G. The impact of missing data on clinical trials: a re-analysis of a placebo controlled trial of Hypericum perforatum (St Johns wort) and sertraline in major depressive disorder. Psychopharmacology (Berl). 2014 May;231(9):1987-99. doi: 10.1007/s00213-013-3344-x. PMID 24232445
- [Derived] Sarris J, Fava M, Schweitzer I, Mischoulon D. St John's wort (Hypericum perforatum) versus sertraline and placebo in major depressive disorder: continuation data from a 26-week RCT. Pharmacopsychiatry. 2012 Nov;45(7):275-8. doi: 10.1055/s-0032-1306348. Epub 2012 May 16. PMID 22592504
- [Derived] Chen JA, Papakostas GI, Youn SJ, Baer L, Clain AJ, Fava M, Mischoulon D. Association between patient beliefs regarding assigned treatment and clinical response: reanalysis of data from the Hypericum Depression Trial Study Group. J Clin Psychiatry. 2011 Dec;72(12):1669-76. doi: 10.4088/JCP.10m06453. Epub 2011 Oct 4. PMID 22053942